CLINICAL TRIAL: NCT00300352
Title: Effect of Folic Acid Treatment in Coronary Artery Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: British Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04.OXB.004
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2007-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Folic acid; Endothelial function
MeSH Terms: conditions — Coronary Artery Disease | interventions — Folic Acid

INTERVENTIONS:
Drug: Folic Acid

SUMMARY:
We seek to examine the effects of folic acid treatment on vascular function in patients with coronary artery disease. Our hypothesis is that folic acid treatment will improve vascular function

DETAILED DESCRIPTION:
Common vascular disease states including diabetes and atherosclerosis are associated with endothelial dysfunction, characterised by reduced bioactivity of nitric oxide (NO). Folates are thought to improve endothelial function,but the mechanism by which this effect occurs is poorly understood. We propose to study the effects of folate supplementation on endothelial function in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of coronary artery disease

Exclusion Criteria:

Recent acute coronary event Renal and/or hepatic dysfunction Metallic implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-05; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Improvement in noninvasive measures of vascular function

SECONDARY OUTCOMES:
Improvement in laboratory measures of vascular function

CONTACTS AND LOCATIONS:
Overall Officials: Keith Channon, MD FRCP, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom